CLINICAL TRIAL: NCT00533182
Title: Influenza in the Non-immunocompromised and Immunocompromised Host
Brief Title: Influenza in People With Normal and Weakened Immune Systems
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 070229; 07-I-0229
Record Dates: First submitted 2007-09-20; First posted 2007-09-21 (Estimated); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Viral Infections; Respiratory Infections
Keywords: Pregnant; Children; Adults; Flu; Infection; Natural History; Influenza Infection
MeSH Terms: conditions — Virus Diseases; Respiratory Tract Infections; Influenza, Human; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole blood, serum, nasal samples

GROUPS / COHORTS (3):
- Immunocompromised: Immunocompromised individuals
- Non-Immunocompromised: Non-immunocompromised individuals
- Pregnant: Pregnant women

SUMMARY:
This study will evaluate how the immune system responds to influenza infection and compare how the infection differs in patients with a weakened immune system versus those with a healthy immune system.

Patients at the NIH Clinical Center who are older than 2 years of age and who are diagnosed with influenza A or B may be eligible for this study. Patients with healthy immune systems and weakened immune systems are included.

Participants answer questions about how they are feeling and have a physical examination to evaluate their symptoms. Blood and nasal fluid are collected on the first day and then every other day for a total of 8 days. Nasal fluid is collected by either inserting a small tube in the nose and washing the nose with salt water and collecting the fluid obtained, or by rubbing the inside of the nose with a swab. Physical examinations are repeated on the days that blood and nasal fluid are collected.

DETAILED DESCRIPTION:
Influenza viruses cause significant morbidity each year, and past epidemics and pandemics have caused significant mortality. The impact influenza has or could have on the increasing number of patients who are immunocompromised due to acute and chronic diseases as well as immunosuppressive therapies is largely unknown. Limited information is available about the innate immune response to influenza and how chronic illness and immunosuppression may affect the immune response to the virus in comparison to that seen in normal hosts.

We will evaluate both immunocompromised and non-immunocompromised (control group) patients from the local community, and the NIH Clinical Center. Patients with known or suspected influenza will be evaluated by recording their symptoms, collecting their blood and nasal specimens, and isolating their viruses. Each patient s infection will be mapped by performing genomic analysis of the viral isolates collected during the patient s infection (which will include analysis of sequences known to confer resistance to antiviral medication), measuring cytokine levels in blood and nasal mucosal samples, and measuring influenza-specific antibody responses. Correlation of these results with clinical symptoms and clinical outcomes will be evaluated. Elucidation of these responses and the genomic changes the virus may undergo during infection and treatment for influenza in both normal and immunocompromised patients may help to better understand the impact influenza has on the overall health of patients, as well as what strategies may be performed to better protect or treat patients during the emergence of a new pandemic.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Greater than or equal to 2 years old
  2. Participant or (LAR) able and willing to complete the consent/assent process and be willing to comply with study procedures
  3. Suspected of having influenza by clinical diagnosis or have a positive clinical diagnostic test for influenza (rapid test molecular test, or culture) within the past 2 months.
  4. Agrees to undergo multiple nasal mucosal sample collections by nasal wash, swab, and/or synthetic absorptive matrix (SAM)
  5. Willing to have blood and nasal samples stored for future use

EXCLUSION CRITERIA:

Participants will not be enrolled in this study if the following criterion applies or is satisfied:

1. Any condition that, in the judgment of the investigator is a contraindication to protocol participation.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with known or suspected influenza infection: NIH Patients, Non-NIH Outpatients, Hospitalized Patients at the Washington Hospital Center, Non-Hospitalized Patients at the Washington Hospital Center. Healthy Pregnant Women (Control): Patients at the Washington Hospital Center
Sampling Method: Probability Sample
Enrollment: 137 (Actual)
Dates: Start 2008-01-03 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2022-08-25 (Actual)

PRIMARY OUTCOMES:
The purpose of this study is to evaluate immunocompromised andnon-immunocompromised individuals who become infected with influenza virus. | 1 year
  To better understand the impact influenza has on the overall health of patients

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J Memoli, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Askonas BA, Lin YL. An influenza specific T-killer clone is restricted to H-2Ld and cross-reacts with Dk region. Immunogenetics. 1982;16(1):83-7. doi: 10.1007/BF00364444. No abstract available. PMID 6981600
- [Background] Couch RB, Kasel JA, Gerin JL, Schulman JL, Kilbourne ED. Induction of partial immunity to influenza by a neuraminidase-specific vaccine. J Infect Dis. 1974 Apr;129(4):411-20. doi: 10.1093/infdis/129.4.411. No abstract available. PMID 4593871
- [Background] McMichael AJ, Gotch FM, Noble GR, Beare PA. Cytotoxic T-cell immunity to influenza. N Engl J Med. 1983 Jul 7;309(1):13-7. doi: 10.1056/NEJM198307073090103. PMID 6602294
- [Derived] Memoli MJ, Athota R, Reed S, Czajkowski L, Bristol T, Proudfoot K, Hagey R, Voell J, Fiorentino C, Ademposi A, Shoham S, Taubenberger JK. The natural history of influenza infection in the severely immunocompromised vs nonimmunocompromised hosts. Clin Infect Dis. 2014 Jan;58(2):214-24. doi: 10.1093/cid/cit725. Epub 2013 Nov 1. PMID 24186906
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2007-I-0229.html